CLINICAL TRIAL: NCT06942208
Title: Iron Revisited: Alternate-Day Oral Iron Supplementation in Endurance, Intermittent, and Power/Strength Athletes
Brief Title: Improving Iron Levels in Female Endurance, Intermittent, and Power/Strength Athletes Aged 16-35
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Mitacs (Industry); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Jane Shearer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB25-0095
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Iron Deficiency
Keywords: iron; iron deficiency; athletic performance; female athlete; iron supplements; ferritin; hemoglobin; gastrointestinal; microbiome; Exercise test; Yeast; Saccharomyces cerevisiae; ferrous sulphate; ferrous sulfate; Body composition; exercise
MeSH Terms: conditions — Iron Deficiencies; Motor Activity | interventions — Iron; ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose iron supplement (Active Comparator): This supplement consists of encapsulated ferrous sulphate (40 mg elemental iron).
  Interventions: Dietary Supplement: Low-dose iron (ferrous sulfate)
- Low dose iron supplement bound to yeast (Experimental): Low dose iron (40 mg elemental iron) in the form of yeast-bound iron, specifically Lalmin® Fe10. This supplement consists of encapsulated ferrous sulphate complexed with inactivated Saccharomyces cerevisiae (nutritional yeast).
  Interventions: Dietary Supplement: Yeast-bound iron (ferrous sulfate)
- High dose iron supplement (Active Comparator): This supplement consists of encapsulated ferrous sulphate (150 mg elemental iron).
  Interventions: Dietary Supplement: High-dose iron (ferrous sulfate)

INTERVENTIONS:
Dietary Supplement: Low-dose iron (ferrous sulfate) — Encapsulated low-dose ferrous sulphate (40mg elemental iron)
  Arms: Low dose iron supplement
Dietary Supplement: Yeast-bound iron (ferrous sulfate) — Encapsulated yeast-bound low-dose ferrous sulphate (40mg elemental iron)
  Arms: Low dose iron supplement bound to yeast
Dietary Supplement: High-dose iron (ferrous sulfate) — Encapsulated high-dose ferrous sulphate (150mg elemental iron)
  Arms: High dose iron supplement

SUMMARY:
The goal of this clinical trial is to learn if different types and doses of oral iron supplements can improve iron levels, athletic performance, and gut health in young female athletes with low iron stores. The main questions it aims to answer are:

* Does a low dose of yeast-bound iron improve iron status better than traditional iron supplements?
* Do the different iron supplements cause fewer or more gastrointestinal (stomach) symptoms?
* How do iron supplements affect exercise performance and gut bacteria?

Researchers will compare three types of iron supplements:

* A low-dose iron supplement (40 mg)
* A low-dose yeast-bound iron supplement (40 mg)
* A high-dose iron supplement (150 mg)

This will help researchers find out which type of supplement is most effective and easiest on the stomach.

Participants will:

* Take one of the three assigned iron supplements every other day for 12 weeks
* Complete fitness tests before and after the study, including cycling and jumping tests
* Give blood samples to measure iron levels
* Provide stool and intestinal samples to study gut bacteria
* Swallow a SIMBA capsule before and after the study to collect a sample from the small intestine
* Complete regular online surveys about sleep, stress, menstrual cycles, and gut symptoms

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate and compare the effects of three oral iron supplementation strategies on iron status, gut microbiota, and athletic performance in young female athletes with suboptimal iron levels. The study compares a low-dose iron supplement, a low-dose yeast-bound iron supplement (Lalmin® Fe10), and a high-dose iron supplement. The primary goal is to identify which iron supplement improves iron status most effectively while minimizing gastrointestinal symptoms and changes to the gut microbiota.

The rationale for the study is based on the high prevalence of iron deficiency among female athletes, especially those involved in endurance and high-intensity sports. Iron plays a key role in oxygen transport, energy production, and recovery, making it essential for optimal athletic performance. However, current supplementation practices often lead to poor compliance due to side effects and low absorption rates. The yeast-bound iron product being tested is hypothesized to improve absorption and tolerability by altering the site of absorption and reducing gastrointestinal distress.

Participants will be biologically female athletes aged 16-35 with suboptimal ferritin (≤50 µg/L), who are competitively trained and meet strict health and fitness criteria. After screening, eligible participants will be randomly assigned to one of three groups and consume their assigned supplement every other day for 12 weeks. Each supplement will be encapsulated to preserve blinding and consistency.

The study involves six in-person visits:

Visit 1 - Screening and Consenting:

Study investigators will reach out electronically or by phone to individuals interested in participating in the study. At this time, participants will be informed about the study and eligibility will be confirmed. Iron status will be assessed using a ferritin blood test from a forearm venipuncture. Participants with suboptimal ferritin levels (≤50 µg/L) will be asked to complete a 3-day food record over the following week on non-consecutive days. This food intake data will be used to determine energy availability to ensure participants meet the minimum requirement of >30 kcal/kg lean body mass. Those who do not meet this requirement will be excluded from further participation.

Visit 2 - Baseline Testing (Week 0):

Eligible participants will return to the lab to undergo baseline testing. This includes another blood draw to confirm iron status, a DXA scan to assess body composition, and a VO2 max test to evaluate aerobic capacity. Participants will also receive a SIMBA capsule, a fecal collection kit, and detailed instructions for home use.

Visit 3 - Baseline Testing (Week 0):

Approximately 48-72 hours after Visit 2, participants will return to the lab for anaerobic performance testing. They will complete a Wingate cycling test and a counter-movement jump test to assess lower-body power and anaerobic fitness. Following this, participants will begin the 12-week supplementation phase of the study.

Nutritional Intervention:

Participants will consume an oral iron supplement every other day for 12 weeks. They will be instructed to take the supplement within 30 minutes of morning training, or upon waking if no training is scheduled. Doses are as follows:

* 40 mg elemental iron (low-dose group)
* 40 mg yeast-bound elemental iron (Lalmin® Fe10 group)
* 150 mg elemental iron (high-dose group)

Each supplement will be delivered in gelatin capsules. Participants will be instructed to avoid coffee, tea, dairy, and dairy alternatives for at least 2 hours after consumption. If a dose is missed, they will resume dosing the next day and continue on an every-other-day schedule. Capsules will be distributed every four weeks. Participants will complete baseline, weekly, and monthly questionnaires through Qualtrics to report gastrointestinal symptoms, stress, sleep, menstrual health, and supplement adherence. These tools include PROMIS-GI, SRSS, GISQ, and others.

Visit 4 - Follow-Up (Week 4):

Participants will return to the lab for a follow-up blood draw to monitor iron status and receive their next 4-week supply of capsules. They will also complete another 3-day food log.

Visit 5 - Post-Intervention Testing (Week 12):

After 12 weeks of supplementation, participants will return for a second VO2 max test. They will return any unused capsules for adherence tracking and be provided instructions for their second SIMBA capsule and fecal sample collection.

Visit 6 - Final Testing (Week 12):

Participants will complete all post-intervention assessments including blood tests, a DXA scan, the Wingate test, the counter-movement jump test, and submission of the second SIMBA capsule and fecal sample. A final 3-day food log will also be collected.

Primary outcomes include changes in markers of iron status (ferritin, hemoglobin, RBC indices). Secondary outcomes include aerobic/anaerobic performance measures, body composition (DXA), substrate metabolism, gut microbiota composition (via fecal and intestinal sampling), and self-reported gastrointestinal symptoms. Safety and tolerability will be monitored at each study visit and through participant self-report.

Data will be analyzed using both traditional statistics (e.g., ANOVA) and machine learning methods for complex 'omics' data. Results will inform better supplementation strategies for female athletes and will be shared through academic publications.

The study will contribute to a greater understanding of iron supplementation strategies that are effective, tolerable, and beneficial to performance and health.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female athlete
* Age 16-35
* At least one year past the age of menarche
* Complete and pass the Get Active Questionnaire (GAQ)
* Suboptimal ferritin levels (≤50 mcg/L)
* Provide informed consent to participate in study
* Activity level based on Participant Classification Framework (McKay et al., 2022)

  * Tier 3: Highly Trained / National Level
  * Tier 4: Elite / International Level
* Energy availability >30 kcal/kg LBM
* Have access to a smartphone, tablet, or computer
* Able to swallow a size-00 capsule (23mm length)

Exclusion Criteria:

* Non-English speaking
* Anemic (hemoglobin <120g/L)
* Antibiotics use within 4 weeks prior to study enrollment
* Regular prebiotic (fiber) or probiotic use within 4 weeks of study enrollment
* Current laxative use
* Are a smoker or use tobacco products
* Consume >21 units of alcohol per week
* Have donated blood in the previous 3 months
* Have a BMI <16 but >30kg/m2
* Are dieting for weight loss or are following a low carbohydrate diet
* Have participated in another clinical trial within the 30 days preceding study enrollment.
* Are taking medications known to affect cardiovascular or metabolic responses to exercise such as beta-blockers, anti-coagulants etc. as assessed by the Principal Investigator.
* Known history of thalassemia or thalassemia trait
* Known inherited bleeding disorder
* Major surgery in the past 3 months
* Chronic use of Salicylates, aspirin, corticosteroids, or nonsteroidal anti-inflammatory drugs
* Have any of the following conditions: renal or gastrointestinal disorders, autoimmune disease, metabolic disease, heart disease, vascular disease, rheumatoid arthritis, diabetes, poor lung function, uncontrolled blood pressure, dizziness, thyroid problems, or any other health conditions that are being treated and deemed to be able to significantly interfere with study intervention and assessment in the opinion of the Principal Investigator and Qualified Investigator
* Have current musculoskeletal injuries that limit exercise capacity
* Self-identifying with any kidney or gastrointestinal issues, metabolic disorders, cardiac conditions, vascular illnesses, rheumatoid arthritis, diabetes, compromised lung function, unregulated blood pressure, episodes of dizziness, thyroid complications, or any other health conditions under treatment that might potentially interfere with the study results
* Orthopaedic issues that limit exercise ability
* Currently/last 3 months taking prescription medications that are known to affect iron absorption (i.e. Antacids/PPIs (e.g., omeprazole), H2 Blockers (e.g., ranitidine), Tetracycline Antibiotics (e.g., doxycycline), Quinolone Antibiotics (e.g., ciprofloxacin), Cholestyramine, Colchicine, Methyldopa.)
* Currently/last 3 months taking iron containing supplements.
* Are pregnant or lactating or planning to become pregnant for the duration of the study. All participants must agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

  * Abstinence or agrees to use contraception if planning to become sexually active
  * Hormonal contraceptives including oral contraceptives, hormone birth control patch
  * Vaginal contraceptive ring, injectable contraceptives, or hormone implant
  * Barrier methods (e.g. condoms with spermicide, diaphragms with spermicide)
  * Intrauterine devices
  * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
  * Vasectomy of partner at least 6 months prior to screening
* Additional exclusion criteria based on use of SIMBA capsules. Following is a summary of SIMBA capsules specific exclusion criteria:

  * Prior gastrointestinal disease, surgery, or radiation treatment which, in the Investigator's opinion, would lead to intestinal structuring or obstruction with a risk of capsule non-excretion, including, e.g. achalasia, eosinophilic esophagitis, any IBD, or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months before the screening visit is acceptable.
  * History of known structural gastrointestinal abnormalities such as structures or fistulas leading to mechanical obstruction
  * Use of any medication in the week prior to the screening study visit, unless part of regular treatment, that could substantially alter gastrointestinal motor function (e.g. opioids, prokinetics, anticholinergics, GLP-1 analogues); laxative use is allowed if it is kept unchanged in the week prior to the study visit. Proton pump inhibitors (PPIs) are allowed provided a wash-out period of 48 hours is respected before swallowing the SIMBA capsules and PPI treatment is resumed only 4 hours thereafter.
  * Organic motility disorder, including gastroparesis, intestinal pseudo-obstruction, systemic sclerosis, Ogilvie's syndrome.
  * History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration
  * Participants schedules for MRI
  * Participants with history of less than 3 bowel movements per week
  * Any prior fecal microbiota transplantation
  * Drug use
* Females of childbearing potential will be asked about their likelihood of being pregnant, based on factors such as recent sexual activity or use of contraception. Their self-reported confirmation of non-pregnancy will be accepted unless they express uncertainty. In cases of doubt, a urine beta-HCG pregnancy test will be required for confirmation.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Iron status blood markers | Baseline
  A forearm venous blood draw (10ml)
  * Ferritin
  * Hemoglobin
Iron status blood markers | 4 weeks
  A forearm venous blood draw (10ml)
  * Ferritin
  * Hemoglobin
Iron status blood markers | 12 weeks
  A forearm venous blood draw (10ml)
  * Ferritin
  * Hemoglobin
Gut microbiota | Baseline
  Effects of the various iron formulations on the gut microbiota using the SIMBA capsule and stool sample analysis.
  Fecal Collection: Participants will provide two stool samples to assess fecal metabolites and gut microbiota composition. Participants will be provided a stool sample collection kit that will allow them to collect the sample in the privacy of their home. The kit will contain all necessary instructions and materials required to perform the collection.
  Gut microbiome Assessment: Participants will ingest a SIMBA capsule pre and post intervention. The capsule captures a small fluid sample from the small intestine, which will be retrieved upon excretion to examine the gut microbiome.
Gut microbiota | 12 weeks
  Effects of the various iron formulations on the gut microbiota using the SIMBA capsule and stool sample analysis.
  Fecal Collection: Participants will provide two stool samples to assess fecal metabolites and gut microbiota composition. Participants will be provided a stool sample collection kit that will allow them to collect the sample in the privacy of their home. The kit will contain all necessary instructions and materials required to perform the collection.
  Gut microbiome Assessment: Participants will ingest a SIMBA capsule pre and post intervention. The capsule captures a small fluid sample from the small intestine, which will be retrieved upon excretion to examine the gut microbiome.

SECONDARY OUTCOMES:
Gut microbiota composition, diversity, and strains recovery | Baseline
  Sample of small intestine microbiota using a SIMBA capsule and fecal sample to determine composition, diversity, and strain recovery.
  Fecal Collection: Participants will provide two stool samples to assess fecal metabolites and gut microbiota composition. Participants will be provided a stool sample collection kit that will allow them to collect the sample in the privacy of their home. The kit will contain all necessary instructions and materials required to perform the collection.
  Gut microbiome Assessment: Participants will ingest a SIMBA capsule pre and post intervention. The capsule captures a small fluid sample from the small intestine, which will be retrieved upon excretion to examine the gut microbiome.
Gut microbiota | 12 weeks
  Sample of small intestine microbiota using a Nimble capsule and fecal sample to determine composition, diversity, and strain.
  Fecal Collection: Participants will provide two stool samples to assess fecal metabolites and gut microbiota composition. Participants will be provided a stool sample collection kit that will allow them to collect the sample in the privacy of their home. The kit will contain all necessary instructions and materials required to perform the collection.
  Gut microbiome Assessment: Participants will ingest a SIMBA capsule pre and post intervention. The capsule captures a small fluid sample from the small intestine, which will be retrieved upon excretion to examine the gut microbiome.
VO2 Max | Baseline
  VO2 max testing on a cycling ergometer to assess peak power output, maximal oxygen consumption, and exercise thresholds.
  Individuals will begin with a 4-minute warm-up of low intensity, then proceed to a progressively increasing cycling challenge until they reach the point of voluntary exhaustion. Breath-by-breath measurement of gas exchange will be captured using open-circuit spirometry at rest, during exercise, and during recovery. Perceptual responses will be recorded during warm-up, every two minutes throughout exercise, and after task failure. Heart rate will be collected using a chest strap and measured throughout exercise. This method is used to evaluate the fitness levels of the participants.
  Metabolic cart measurements: Participants will wear a mask connected to a breath-by-breath metabolic cart to measure expired gases and minute ventilation. This equipment will continuously monitor the expired concentrations of O2 and CO2.
VO2 Max | 12 weeks
  VO2 max testing on a cycling ergometer to assess peak power output, maximal oxygen consumption, and exercise thresholds.
  Individuals will begin with a 4-minute warm-up of low intensity, then proceed to a progressively increasing cycling challenge until they reach the point of voluntary exhaustion. Breath-by-breath measurement of gas exchange will be captured using open-circuit spirometry at rest, during exercise, and during recovery. Perceptual responses will be recorded during warm-up, every two minutes throughout exercise, and after task failure. Heart rate will be collected using a chest strap and measured throughout exercise. This method is used to evaluate the fitness levels of the participants.
  Metabolic cart measurements: Participants will wear a mask connected to a breath-by-breath metabolic cart to measure expired gases and minute ventilation. This equipment will continuously monitor the expired concentrations of O2 and CO2.
Wingate | Baseline
  Wingate test completed on cycle ergometer to determine peak power output and fatigue index.
  During this test, participants will use a cycle ergometer. After a five-minute warm-up at low intensity, participants will pedal at maximum effort against a set resistance (7.5%) for 30 seconds, based on their body weight. Peak power will be assessed as well as other key performance metrics.
Wingate | 12 weeks
  Wingate test completed on cycle ergometer to determine peak power output and fatigue index.
  During this test, participants will use a cycle ergometer. After a five-minute warm-up at low intensity, participants will pedal at maximum effort against a set resistance (7.5%) for 30 seconds, based on their body weight. Peak power will be assessed as well as other key performance metrics.
Counter-movement jump test | Baseline
  Three sets of fifteen consecutive counter-movement jumps on a force plate to assess lower body power and explosive strength. Participants will stand with their hands on their hips, bend their knees rapidly to lower into a squat position, followed by an explosive vertical jump. They will be allowed two seconds between each jump and 60 seconds between each set. Testing will occur before (baseline) and after supplementation (2 times total).
Counter-movement jump test | 12 weeks
  Three sets of fifteen consecutive counter-movement jumps on a force plate to assess lower body power and explosive strength. Participants will stand with their hands on their hips, bend their knees rapidly to lower into a squat position, followed by an explosive vertical jump. They will be allowed two seconds between each jump and 60 seconds between each set. Testing will occur before (baseline) and after supplementation (2 times total).
Body composition | Baseline
  The DXA procedure uses a small amount of x-ray radiation to determine the amount of fat, bone, and muscle mass an individual has in his/her body.
Body composition | 12 weeks
  The DXA procedure uses a small amount of x-ray radiation to determine the amount of fat, bone, and muscle mass an individual has in his/her body.
Gastrointestinal Health | Weekly from baseline to 12 weeks
  PROMIS and GI Symptom Rating Scale questionnaires to assess gastrointestinal symptoms.
Menstrual cycle | Baseline
  MDOT questionnaire to assess menstrual cycle.
Menstrual cycle | baseline
  Menstrual Bleeding questionnaire to assess menstrual cycle.
Menstrual cycle | 4 weeks
  Menstrual Bleeding questionnaire to assess menstrual cycle.
Menstrual cycle | 8 weeks
  Menstrual Bleeding questionnaire to assess menstrual cycle.
Menstrual cycle | 12 weeks
  Menstrual Bleeding questionnaire to assess menstrual cycle.
Short Stress and Recovery Scale (SSRS) | Completed weekly from baseline to 12 weeks
  Short Stress and Recovery Scale (SSRS) to assess recovery and stress; higher scores under each domain indicate higher levels of stress or recovery, respectively
Activity Readiness | Baseline
  Get Active Questionnaire to assess readiness for exercise.
Sleep | Baseline
  Epworth Sleepiness Scale (ES) to assess sleep; possible range 0-24; higher scores indicate higher levels of sleepiness
Sleep | 4 weeks
  Epworth Sleepiness Scale (ES) to assess sleep; possible range 0-24; higher scores indicate higher levels of sleepiness
Sleep | 12 weeks
  Epworth Sleepiness Scale (ES) to assess sleep; possible range 0-24; higher scores indicate higher levels of sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Jane Shearer, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantopoulos K. Oral iron supplementation: new formulations, old questions. Haematologica. 2024 Sep 1;109(9):2790-2801. doi: 10.3324/haematol.2024.284967. PMID 38618666
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513
- [Background] McKay AKA, Sim M, Moretti D, Hall R, Stellingwerff T, Burden RJ, Peeling P. Methodological Considerations for Investigating Iron Status and Regulation in Exercise and Sport Science Studies. Int J Sport Nutr Exerc Metab. 2022 Apr 1;32(5):359-370. doi: 10.1123/ijsnem.2021-0343. Print 2022 Sep 1. PMID 35365588
- [Background] McCormick R, Moretti D, McKay AKA, Laarakkers CM, Vanswelm R, Trinder D, Cox GR, Zimmerman MB, Sim M, Goodman C, Dawson B, Peeling P. The Impact of Morning versus Afternoon Exercise on Iron Absorption in Athletes. Med Sci Sports Exerc. 2019 Oct;51(10):2147-2155. doi: 10.1249/MSS.0000000000002026. PMID 31058762
- [Background] Low MS, Speedy J, Styles CE, De-Regil LM, Pasricha SR. Daily iron supplementation for improving anaemia, iron status and health in menstruating women. Cochrane Database Syst Rev. 2016 Apr 18;4(4):CD009747. doi: 10.1002/14651858.CD009747.pub2. PMID 27087396
- [Background] Erdman KA, Fung TS, Doyle-Baker PK, Verhoef MJ, Reimer RA. Dietary supplementation of high-performance Canadian athletes by age and gender. Clin J Sport Med. 2007 Nov;17(6):458-64. doi: 10.1097/JSM.0b013e31815aed33. PMID 17993788
- [Background] Cordova A, Mielgo-Ayuso J, Fernandez-Lazaro CI, Caballero-Garcia A, Roche E, Fernandez-Lazaro D. Effect of Iron Supplementation on the Modulation of Iron Metabolism, Muscle Damage Biomarkers and Cortisol in Professional Cyclists. Nutrients. 2019 Feb 27;11(3):500. doi: 10.3390/nu11030500. PMID 30818782
- [Background] Attwell C, McKay A, Sim M, Dugan C, Nicholas J, Hopper L, Peeling P. Timing is everything, but does it really matter? Impact of 8-weeks morning versus evening iron supplementation in ballet and contemporary dancers. Eur J Sport Sci. 2023 Dec;23(12):2275-2282. doi: 10.1080/17461391.2023.2224285. Epub 2023 Jul 10. PMID 37291690